CLINICAL TRIAL: NCT01992133
Title: The Effects of Vitamin D Supplementation on Blood Glucose and Markers of Metabolic Syndrome in Women With Vitamin D Deficiency and Previous Gestational Diabetes Mellitus
Brief Title: Effects of Vitamin D Supplementation on Glucose Metabolism in Women With Former Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RCSI & UCD Malaysia Campus (Other)
Responsible Party: Principal Investigator, Toh-Peng Yeow, Assoc Professor of Medicine, RCSI & UCD Malaysia Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRR-10-679-6202
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Vitamin D Deficiency
Keywords: Former gestational Diabetes; Vitamin D deficiency; insulin resistance; beta cell function
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 at 4000 iu per day for 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): matching placebo- capsules containing soya oil at 4 capsules a day for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Arms: Vitamin D3
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Gestational Diabetes Mellitus (GDM) and vitamin D deficiency are related to insulin resistance and impaired beta-cell function, with heightened risk for future development of diabetes. The investigators hypothesize that vitamin D supplementation to women with previous gestational diabetes may improve glucose metabolism.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is a state of glucose intolerance occurring during pregnancy and is related to both resistance to peripheral action of insulin and impairment of beta (β)-cell function. Its transient presence during pregnancy alerts to a heightened risk of diabetes in the future. About 10-50% of women with GDM develop diabetes mellitus later on in life. Data from Malaysia found that 50% of GDM women had developed diabetes at an interval of five to seven years post index pregnancy. Therefore, it is paramount that the investigators identify effective measures to prevent diabetes progression in this high-risk group.

Vitamin D deficiency has been shown to be associated with insulin resistance and impaired pancreatic function. Vitamin D deficiency is more prevalent in women with GDM and low vitamin D levels correlate with insulin resistance.

Interventional studies using vitamin D supplement in an attempt to modify glucose metabolism have yielded mixed results. This may be partly due to variable doses of supplementation used, short duration of follow up and inappropriate target group. A very short duration of less than seven days of supplementation may not be sufficient to demonstrate the potential beneficial effects. Previous studies suggested vitamin D replacement improved glucose metabolism in selected populations only. Benefit was seen in subjects with impaired fasting glucose but not in normal volunteers, nor in patients with established chronic diabetes. It is possible that vitamin D can help with early stage of disturbance in glucose handling, but is unable to augment insulin secretion in subjects with chronic diabetes and exhausted pancreatic function. Lack of adequate dosing may have also accounted for the failure of many previous studies to demonstrate beneficial effects of vitamin D replacement. Adequate vitamin D supplementation would ideally raise blood 25-hydroxyvitamin D (25(OH)D) levels above 80nmol/L because diabetes risk is lowest at this vitamin D level. Supplementation with 4000IU of vitamin D3 per day in a population of South Asian women with proven vitamin D deficiency safely restored the vitamin D level and improved insulin resistance.

Very little is known about the relationship between vitamin D status and glucose metabolism in women with former GDM. This study aimed to evaluate the effect of adequate vitamin D supplementation on insulin sensitivity, pancreatic β-cell function and markers of cardio-metabolic risk in Malaysian women with former GDM and vitamin D insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Women with Gestational Diabetes (GDM) on the most recent pregnancy- between 6 and 48 months post partum at time of recruitment to study
* Previous GDM defined as-Fasting plasma glucose ≥ 7.0 mmol/l or 2-h plasma glucose ≥ 7.8 mmol/l on 75g OGTT performed during gestation OR As determined by treating physician during index pregnancy
* With no plan to conceive again within the 6 months of study duration
* With 75g OGTT at study baseline confirming either Normal respond, Impaired Fasting Glucose (IFG) or Impaired Glucose Tolerance (IGT)
* Vitamin D deficiency at baseline - defined as Plasma 25-(OH) D concentration of between 15 and 50nmol/L

Exclusion Criteria:

* Pregnancy or Breast feeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in glucose metabolism as assessed by change in Insulin sensitivity index as calculated by HOMA -IR28 | 6 months

SECONDARY OUTCOMES:
Change in Insulin Sensitivity index as calculated by Oral Glucose Insulin Sensitivity Index (OGIS) | 6 months
Change in plasma 25-OH- Vitamin D level pre and post replacement | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Toh Peng Yeow, MB BCH BAO, FRCP(Edin), Principal Investigator — Penang Medical College, 4 Jalan Sepoy Lines, 11450, Penang, Malaysia
Locations (1):
- Penang Medical College, George Town, Malaysia